CLINICAL TRIAL: NCT07255131
Title: The Effectiveness and Efficacy of an Online Group Cognitive Behavioral Psychotherapy in Patients With Cystic Fibrosis and Caregivers in Comparison to Control Groups by the Hellenic Cystic Fibrosis Association A Randomized Controlled Trial
Brief Title: The Effectiveness and Efficacy of an Online Cognitive Behavioral Psychotherapeutic Program
Acronym: RAKITZIHCFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rakitzi, Stavroula (Other)
Responsible Party: Principal Investigator, Dr. Stavroula Rakitzi, PhD, Clinical psychologist and cognitive behavioral psychotherapist, Rakitzi, Stavroula
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAKITZI CYSTIC FIBROSIS; HELLENIC CYSTIC FIBROSIS ASSOC (Other: HELLENIC CYSTIC FIBROSIS ASSOCIATION & DR. STAVROULA RAKITZI)
Record Dates: First submitted 2025-09-26; First posted 2025-11-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; Anxiety Chronic; Anxiety; Functional Outcome; Recovery; Obsessive Compulsive Disorders; Assertiveness
Keywords: Cystic Fibrosis; Group cognitive behavioral psychotherapy
MeSH Terms: conditions — Anxiety Disorders; Compulsive Personality Disorder; Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: A therapy group with patients with cystic fibrosis will be compared with a control group with patients with cystic fibrosis. A therapy group with caregivers will be compared with a control group with cqaregivers
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Therapy group A patients with Cystic Fibrosis (Experimental): Participation on an online group cognitive behavioral psychotherapy via Zoom in 13 sessions.
  3 participants
  Interventions: Behavioral: Group A An online group cognitive behavioral psychotherapy in 13 sessions via Zoom
- Control group B Patients with cystic fibrosis (Active Comparator): Participation on an online group supportive psychotherapy via Zoom in 13 sessions.
  2 participants
  Interventions: Behavioral: Group B An online group supportive psychotherapy in 13 sessions via Zoom
- Therapy group C caregivers of patients with cystic fibrosis (Experimental): Participation on an online group cognitive behavioral psychotherapy via Zoom in 13 sessions.
  2 participants
  Interventions: Behavioral: Group C An online group cognitive behavioral psychotherapy in 13 sessions via Zoom
- Contol group D caregivers of patients with cystic fibrosis (Active Comparator): Participation on an online group supportive psychotherapy via Zoom in 13 sessions.
  2 participants
  Interventions: Behavioral: Group D An online group supportive psychotherapy in 13 sessions via Zoom

INTERVENTIONS:
Behavioral: Group A An online group cognitive behavioral psychotherapy in 13 sessions via Zoom — An online group cognitive behavioral psychotherapy will be offered via Zoom in 13 sessions to the therapy Group A, to patients with cystic fibrosis
  Other Names: Experimental
  Arms: Therapy group A patients with Cystic Fibrosis
Behavioral: Group B An online group supportive psychotherapy in 13 sessions via Zoom — An online group supportive psychotherapy will be offered via Zoom in 13 sessions to the control group Group B, to patients with cystic fibrosis
  Other Names: Active comparator
  Arms: Control group B Patients with cystic fibrosis
Behavioral: Group C An online group cognitive behavioral psychotherapy in 13 sessions via Zoom — An online group cognitive behavioral psychotherapy will be offered via Zoom in 13 sessions to the therapy group C, to caregivers of patients with cystic fibrosis
  Other Names: Experimental
  Arms: Therapy group C caregivers of patients with cystic fibrosis
Behavioral: Group D An online group supportive psychotherapy in 13 sessions via Zoom — An online group supportive psychotherapy will be offered via Zoom in 13 sessions to the control Group D, to caregivers of patients with cystic fibrosis
  Other Names: Active comparator
  Arms: Contol group D caregivers of patients with cystic fibrosis

SUMMARY:
An online group cognitive behavioral psychotherapeutic program will be offered to patients with cystic fibrosis and to caregivers by the Hellenic Cystic Fibrosis Association. These 2 above therapy groups will be compared with control groups in a randomized controlled trial

DETAILED DESCRIPTION:
A therapy group of patients with cystic fibrosis, who participate on the online group cognitive behavioral psychotherapeutic program will be compared with a control group of patients with cystic fibrosis, who participate in an online group supportive psychotherapeutic program. Both of the groups participate on 13 sessions once a week.

A therapy group of caregivers, who participate on the online group cognitive behavioral psychotherapeutic program will be compared with a control group of caregivers, who participate in an online group supportive psychotherapeutic program. Both of the groups participate on 13 sessions once a week.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Members of the Hellenic Cystic Fibrosis Association
* Willingness to participate on 13 sessions via Zoom

Exclusion Criteria:

* Age over 70
* Not members of the Hellenic Cystic Fibrosis Association
* Not able to participate on 13 sessions via Zoom

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
SCL-90-R | Preintervention
  It evaluates psychopathology. T>60 means psychopathology. Low scores better
SCL-90-R | Immediately after the intervention
  It evaluates psychopathology. T>60 means psychopathology. Low scores better
SCL-90-R | Follow-up up to 24 weeks
  It evaluates psychopathology. T>60 means psychopathology. Low scores better
SRSDA | Preintervention
  It measures Depression. Minimum 0 Maximum over 14. Low scores better
SRSDA | Immediately after intervention
  It measures Depression. Minimum 0 Maximum over 14. Low scores better
SRSDA | Follow-up up to 24 weeks
  It measures Depression. Minimum 0 Maximum over 14. Low scores better
SRSDA | Preintervention
  It measures anxiety. Minimum 0 Maximum over 10. Low scores better
SRSDA | Immediately after intervention
  It measures anxiety. Minimum 0 Maximum over 10. Low scores better
SRSDA | Follow-up up to 24 weeks
  It measures anxiety. Minimum 0 Maximum over 10. Low scores better
U Uncertainty questionnaire | Preintervention
  It evaluates social skills and assertiveness.: fear of criticism (psychopathology in >35), fear of contact (psychopathology in >41) , assertiveness (psychopathology in <26) , difficulty of saying no (psychopathology in >28) , guilt and decency (psychopathology in >9)
U Uncertainty questionnaire | Immediately after the intervention
  It evaluates social skills and assertiveness.: fear of criticism (psychopathology in >35), fear of contact (psychopathology in >41) , assertiveness (psychopathology in <26) , difficulty of saying no (psychopathology in >28) , guilt and decency (psychopathology in >9)
U Uncertainty questionnaire | Follow up up to 24 weeks
  It evaluates social skills and assertiveness.: fear of criticism (psychopathology in >35), fear of contact (psychopathology in >41) , assertiveness (psychopathology in <26) , difficulty of saying no (psychopathology in >28) , guilt and decency (psychopathology in >9)
Hamilton Depression Scale | Preintervention
  It measures depression. Minimum 0, maximum 23. Low scores better.
Hamilton Depression Scale | Immediately after the intervention
  It measures depression. Minimum 0, maximum 23. Low scores better.
Hamilton Depression Scale | Follow up up to 24 weeks
  It measures depression. Minimum 0, maximum 23. Low scores better.
WHODAS total | Preintervention
  It measures functional outcome. Minimum 0, maximum 100. low scores better.
WHODAS total | Immediately after the intervention
  It measures functional outcome. Minimum 0, maximum 100. low scores better.
WHODAS total | Follow up up to 24 weeks
  It measures functional outcome. Minimum 0, maximum 100. low scores better.
RAS-DS total | Preintervention
  Recovery. It measures recovery. Minimum 0, maximum 152. High scores better.
RAS-DS total | Immediately after intervention
  Recovery. It measures recovery. Minimum 0, maximum 152. High scores better.
RAS-DS total | Follow up up to 24 weeks
  Recovery. It measures recovery. Minimum 0, maximum 152. High scores better.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Stavroula Rakitzi, Study Chair — Private Practice
Locations (1):
- Private practice, ILISION 34 15771 Athens Greece, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
This is our first effectiveness and efficacy study regarding the comparison of the online group cognitive behavioral program for patients with cystic fibrosis and caregivers in comparison to control groups

REFERENCES:
- [Background] Rakitzi, S., Spinou, A., & Giannaki, K. (2025). The effectiveness of an online-group cognitive behavioral psychotherapy in Hellenic Cystic Fibrosis Association for patients and caregivers. Journal of rational emotive and cognitive behavior therapy. DOI: 10.1007/s10942-025-00611-3
- [Background] Rakitzi, S. (2023). Clinical psychology and cognitive behavioral psychotherapy. Recovery in mental health. Springer.
- [Background] Mayr, S., Erdfelder, E., Buchner, A., & Faul, F. (2007). A short tutorial of G-Power. Tutorials in Quantitative Methods in Psychology, 3(2), 51-59.
- [Background] Koumpouros, Y., Papageorgiou, E., Sakellari, E., Prapas, X., Perifanou, D., & Lagiou, A. (2018). Adaptation and psychometric properties' evaluation of the Greek version of WHODAS 2.0. Pilot application in Greek elderly population. Health Services and Outcomes Research Methodology, 18(1), 63-74. https://doi.org/10.1007/s10742-017-0176-x.
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Hancock N, Scanlan JN, Honey A, Bundy AC, O'Shea K. Recovery Assessment Scale - Domains and Stages (RAS-DS): Its feasibility and outcome measurement capacity. Aust N Z J Psychiatry. 2015 Jul;49(7):624-33. doi: 10.1177/0004867414564084. Epub 2014 Dec 19. PMID 25526940
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Fountoulakis KN, Iacovides A, Kleanthous S, Samolis S, Gougoulias K, St Kaprinis G, Bech P. The Greek translation of the symptoms rating scale for depression and anxiety: preliminary results of the validation study. BMC Psychiatry. 2003 Dec 10;3:21. doi: 10.1186/1471-244X-3-21. PMID 14667249
- [Background] Fiedler, P. (2005). Verhaltenstherapie in Gruppen. Beltz.
- [Background] Cohen, J. (1988). Statistical Power Analyses for the Behavioural Sciences. Erlbaum.
- [Background] Bech, P. (1993). Rating scales for Psychopathology, Health Status and Quality of Life. Springer-Verlag.
- [Background] Αntoniou, V., Εfthimiou, Κ., & Μilona, Κ.(2015). Social anxiety and assertiveness. A structured group cognitive behavioral program. IETHS.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT07255131/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT07255131/ICF_001.pdf